CLINICAL TRIAL: NCT04740177
Title: Epidemiology of Congenital Heart Disease in France : EPIDEMIO-CHD
Brief Title: Epidemiology of Congenital Heart Disease in France
Acronym: EPIDEMIO-CHD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: National Reference Center for Complex Congenital Heart Disease, Marie-Lannelongue Medical and Surgical Center, Le Plessis Robinson (Unknown); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0119
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-01

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; Paediatric cardiology; Epidemiology; M3C network
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart disease (CHD) is the leading cause of birth defects, with an incidence of 0.8%. Since the 1980s, France has been a pioneer in neonatal CHD surgery (Pr. Fontan, Pr. Lecomte, Pr. Serraf, etc.), in prenatal diagnosis, and in interventional cardiac catheterization.

Actually, first children operated for complex CHD have reached adulthood and a new epidemiology of CHD is emerging. Currently, one of the public health challenges is the need to maintain appropriate follow-up and to avoid disruption of care during the transition from adolescence to adulthood. Thus, the national health authorities (DGOS) recently certified a national network of expert centers for complex CHD (M3C).

In addition, under the leadership of the French Society of Cardiology, the sub-specialty of Pediatric and Congenital Cardiology has been recognized.

However, while North American and North European countries have published their updated data on the main indicators of CHD morbidity and mortality, no study has reported epidemiology of CHD in France.

Currently, available data are approximate, estimating that 200,000 children and 250,000 adults would be living in France with a CHD. Nevertheless, no information is available on hospitalizations, type of CHD, their follow-up, possible disruption in care, and morbidity and mortality in patients with CHD in France. This epidemiological study will use the national health insurance hospital database to answer these questions.

DETAILED DESCRIPTION:
Retrospective epidemiological study based on the national health insurance hospital database from 2010 to 2020 (10 years):

Main objective:

• To assess the prevalence of patients with CHD hospitalized in France over 10 years.

Secondary objectives: asess over the same period:

* Overall mortality rate according to the CHD classification and the geographic area
* Overall morbidity rate, according to the CHD classification and the geographic area
* Overall cardiac surgery-related mortality rate (cardiac surgery and other surgery), according to the CHD classification (adjusted for the severity of the CHD and the surgical procedure) and to geographic area
* Overall cardiac catheter-related mortality rate, according to the CHD classification (adjusted for the severity of the CHD and the catheterization procedure) and to geographic area
* CHD follow-up within and outside the national M3C network
* Periods of loss of cardiological follow-up (within or outside the M3C network, in hospital or in town)
* Obstetrical data for women (parity, pregnancy)
* The existence of a prenatal diagnosis (yes / no and the term of pregnancy at the time of diagnosis of CHD)

ELIGIBILITY:
Inclusion criteria:

- Patient (of any age) with a CHD as defined by the international ACC-CHD classification and listed in the ICD10 classification, hospitalized from 01/01/2010 to 12/31/2019 in a French tertiary care hospital from the M3C network.

Exclusion criteria:

- Patient with non-malformative genetic heart disease (cardiomyopathy, hereditary rhythmic disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with congenital heart disease (CHD)
Sampling Method: Non-Probability Sample
Enrollment: 450000 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of patients with CHD hospitalized in France | 10 years
  Rate of patients with CHD hospitalized in France

SECONDARY OUTCOMES:
Rate of mortality in patients with CHD | 10 years
  Rate of mortality in patients with CHD
Rate of cardiac surgery-related mortality in patients with CHD | 10 years
  Rate of cardiac surgery-related mortality in patients with CHD
Rate of cardiac catheter-related mortality in patients with CHD | 10 years
  Rate of cardiac catheter-related mortality in patients with CHD
Rate of CHD patient's loss to follow-up within and outside the national M3C network | 10 years
  Rate of CHD patient's loss to follow-up within and outside the national M3C network
Rate of CHD prenatal diagnosis | 10 years
  Rate of CHD prenatal diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD-PhD, Study Director — UH MONTPELLIER; Sarah Cohen, Principal Investigator — • Centre Médico-Chirurgical Marie-Lannelongue, Le Plessis Robinson; Jean-Benoit Thambo, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC